CLINICAL TRIAL: NCT04662138
Title: Safety and Efficacy of Directly Acting Antiviral Agents in Genotype 4 Hepatitis C Virus Relapse Among Egyptian Patients
Brief Title: Safety and Efficacy of Different Antiviral Regimens for Hepatitis C Virus Relapse
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Other Study IDs: 0304769
Record Dates: First submitted 2020-12-04; First posted 2020-12-10 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-08

CONDITIONS: Hepatitis C; Relapse; Antivirals
MeSH Terms: conditions — Hepatitis C; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: directly acting antivirals — Different regimens given for genotype 4 relapse: Sofosbuvir/velpatasvir/voxilaprevir ±ribavirin; sofosbuvir/velpatasvir ±ribavirin; ombitasvir/paritaprevir/ritonavir+ ribavirin

SUMMARY:
The primary goal of hepatitis C virus (HCV) Direct Acting Antivirals (DAAs) is to achieve undetectable HCV RNA in the blood. A response that should be maintained for at least 12 weeks from completion of therapy. This is called sustained virological response (SVR) which corresponds to cure of HCV infection as risk of later relapse is very small. SVR is important to achieve improvement in liver necroinflammation and fibrosis and to decrease complications of cirrhosis.

Failing to achieve SVR after treatment requires another regimen for these experienced patients.

Real-world data are always needed to evaluate and improve our practices. Here investigators aim to assess tolerability and efficacy of different regimens used for management of genotype 4 HCV relapse.

ELIGIBILITY:
Inclusion Criteria:

* all patients with HCV relapse after sofosbuvir plus either Non-structural protein 5 A (NS5A) or protease inhibitor.

Exclusion Criteria:

* No exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with HCV relapse after sofosbuvir plus either NS5A or protease inhibitor who will start another HCV treatment at Alexandria University Viral Hepatitis Treatment Unit or Alexandria University Liver Clinics in the period from 24/8/2020 to 23/8/2021.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-08-24 (Actual); Primary Completion 2022-05-28 (Estimated); Study Completion 2022-05-28 (Estimated)

PRIMARY OUTCOMES:
Sustained virological response | 12 weeks after completion of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria University., Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes